CLINICAL TRIAL: NCT03787290
Title: Examining Immune-Based Mechanisms of Action for Mild-Intensity Whole Body Hyperthermia (WBH) in the Treatment of Major Depressive Disorder
Brief Title: Mild-Intensity Whole Body Hyperthermia (WBH) for Major Depressive Disorder
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: we were not able to get the study drug due to covid
Sponsor: Massachusetts General Hospital (Other)
Collaborators: heckel medizintechnik GmbH (Unknown)
Responsible Party: Principal Investigator, David Mischoulon, MD, PhD, Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020P002424
Record Dates: First submitted 2018-10-27; First posted 2018-12-26 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Major Depressive Disorder
Keywords: hyperthermia; whole-body hyperthermia; depression; major depressive disorder; cytokine; inflammation; immunological; mechanism of action; tocilizumab
MeSH Terms: conditions — Depressive Disorder, Major; Hyperthermia; Depression; Inflammation | interventions — tocilizumab; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomization will be conducted by randomly permuted blocks of 4. The randomization schedule will be created by a statistician who has no other role in the study data collection or analysis. The randomization schedule will be sent directly from the statistician to the Research Pharmacy which will maintain the list. Qualifying study subjects will be assigned the next sequential treatment assignment on the randomization schedule, in the order they are randomized. Participants will be randomized on a 1-to-1 allocation to one of two study arms: 1) tocilizumab followed by whole body hyperthermia (WBH); or 2) placebo followed by whole body hyperthermia (WBH). At the time of randomization, the study coordinator will contact the Research Pharmacy to complete the coded treatment assignment described below.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomization list maintained by the Research Pharmacy will contain the treatment assignment, along with a letter code (A or B) corresponding to the two treatment groups. During the study period and continuing until the major hypotheses have been tested and reported, the correspondence of letter-coded treatment assignment to actual treatment (tocilizumab or placebo) will be known only by pharmacy staff. The study principal investigator (PI), study coordinators, clinicians conducting outcome assessments, and study statistician, as well as research assistants interacting with patients or entering study data and laboratory technicians performing/reporting biomarker assays, will have no access to any subject's treatment assignment. Only after the study statistician has completed and reported analyses by coded treatment assignment for the study aims articulated in this protocol will the correspondence between letter codes and actual treatment be revealed to study personnel.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Tocilizumab (Experimental): Participants will receive tocilizumab followed by whole-body hyperthermia
  Interventions: Drug: Tocilizumab; Device: Whole-Body Hyperthermia
- Placebo (Active Comparator): Participants will receive a placebo followed by whole-body hyperthermia
  Interventions: Drug: Placebo; Device: Whole-Body Hyperthermia

INTERVENTIONS:
Drug: Tocilizumab — participants will receive a single subcutaneous injection of tocilizumab (162 mg)
  Arms: Tocilizumab
Drug: Placebo — participants will receive a single subcutaneous injection of saline
  Other Names: Saline
  Arms: Placebo
Device: Whole-Body Hyperthermia — subjects' core temperature will be increased to 38.5 degrees Celsius (typically 60-120 minutes) then they will begin a 60-minute cool-down phase
  Other Names: Heckel HT3000

SUMMARY:
Overall, the objective of this pilot study is to utilize the IL-6 receptor antagonist tocilizumab to prospectively evaluate the role of IL-6 in the antidepressant and immunological effects of whole body hyperthermia (WBH). The study seeks to replicate findings thus far that WBH has an antidepressant effect by administering the intervention at a site not involved in studies to date. Moreover, the current proposal may help the investigators better understand the role of IL-6 in the pathogenesis and treatment of depression which might point to novel immune-based interventions for Major Depressive Disorder (MDD). Finally, the current proposal holds promise for better understanding of a novel treatment for MDD, which is among the leading causes of health-related disability in the world.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is among the leading causes of overall global disease burden. Much of this burden derives from the fact that currently available pharmacologic modalities suffer from important shortcomings, including limited efficacy, delayed onset of action, and significant side effects that impair quality of life and promote treatment non-adherence and/or discontinuation. These factors provide ample incentive to continue the search for novel antidepressant methodologies that might maximize the benefits of these newer treatment modalities while minimizing their limitations. It is within this context that discoveries regarding the use of whole body hyperthermia (WBH) are of significant potential clinical relevance. The investigators' studies to date suggest that WBH produces a rapid and sustained antidepressant response with an extremely favorable side effect profile in medically-healthy patients with MDD. To follow up on evidence of the antidepressant effect of hyperthermia observed in animal models, the investigators conducted an open trial of WBH in humans. In 16 medically-healthy adults with MDD, the investigators found that a single session of WBH induced a rapid, robust and sustained reduction in depressive symptom scores (Hanusch et al. 2013). Thirteen of the study participants received no other pharmacologic or psychotherapeutic intervention during the study period (pre-treatment and 5 days post-treatment), whereas 3 participants were receiving a stable dose prior to treatment with a selective serotonin reuptake inhibitor (SSRI) antidepressant (with no change in dosage during the study period). Interestingly, when looked at separately, WBH appeared to have no effect in these 3 individuals, and, in fact, worsened depressive symptoms in one of them. These findings are consonant with animal data from the investigators' group demonstrating that therapeutic doses of an SSRI (citalopram 20 mg/kg) obviated the antidepressant-like effects of WBH (Hale et al. 2017).

The investigators' group followed-up positive findings from this initial open trial with a randomized, double-blind, sham-controlled study of WBH. Confirming the investigators primary study hypothesis, participants in the active WBH group showed significantly reduced Hamilton Depression Rating Scale (HDRS) scores at one week post-treatment when compared to participants in the sham group. A similar advantage for active WBH at one week post-treatment was apparent based on self-reported Inventory of Depressive Symptomatology Self-Report (IDS-SR) scores which indicated that active WBH separated from sham beginning on day 3 post-treatment. Contrary to the investigators' a priori hypothesis, the antidepressant effect of active WBH remained apparent out to 6 weeks post treatment when compared to sham. Based on HDRS scores, 60% (9 of 15) of the active WBH group met criteria for response and 40% (6 of 15) met criteria for remission during at least one post-intervention assessment, compared with 7% (1 of 14) and 0% respectively for sham. Rates of adverse events were very low in both WBH and sham groups, with no differences between groups, except for increased adverse events at post-intervention week two in the sham group (Janssen et al. 2016).

With regards to the immunosuppressive effects of WBH, much of the investigators' prior work has focused on the role of inflammation in the etiology and treatment of MDD. Given this, in the investigators' initial randomized, sham-controlled, double-blind trial of WBH they examined the impact of WBH on inflammatory cytokines (tumor necrosis factor [TNF], interleukin (IL)-6, IL-1-beta). Based on extensive data from the investigators' group and many others indicating that the cytokines TNF and IL-6 have depressogenic potential and are elevated in MDD, the investigators sought to test the hypothesis that WBH would reduce plasma concentrations of these cytokines and that these reductions would be associated with improved mood. However, when compared to sham, WBH produced a striking acute increase in IL-6 that resolved completely by one-week post-intervention, while having no acute or chronic effect on TNF.

Because IL-6 can come from multiple cell types in the body, and may have more of a pro-inflammatory vs. anti-inflammatory effect depending on whether it comes from immune cells (pro-inflammatory) or other tissues (i.e. adipocytes, muscle fibers, skin cells) (anti-inflammatory), the investigators measured plasma neopterin concentrations prior to, and following, the study interventions and at post-intervention weeks 1 and 4 simultaneous with the measurement of IL-6.

The investigators next explored whether acute changes in IL-6 and/or neopterin were associated with the antidepressant effects of WBH. The investigators found that acute increases in both IL-6 and neopterin in response to WBH were associated with reduced self-reported depressive symptoms one week following the treatment. Smaller but similar associations were observed between this immune signal and reductions in clinician-rated HDRS scores at one-week post-treatment. Increased IL-6 and neopterin in response to WBH were also associated with increased positive emotion from beginning to conclusion of the procedure.

Overall, the objective of this pilot study is to utilize the IL-6 receptor antagonist tocilizumab to prospectively evaluate the role of IL-6 in the antidepressant and immunological effects of WBH. The study will seek to replicate findings thus far that WBH has an antidepressant effect by administering the intervention at a site not involved in studies to date. Moreover, the current proposal may help the investigators better understand the role of IL-6 in the pathogenesis and treatment of depression which might point to novel immune-based interventions for MDD . Finally, the current proposal holds promise for better understanding a novel treatment for MDD, which is among the leading causes of health-related disability in the world.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide informed consent for study participation.
2. Males and females between the age of 18 and 65 years.
3. Have a current primary psychiatric diagnosis of major depressive disorder (MDD) of at least 4 weeks duration, as defined by DSM-5 criteria using the MINI v.7.0.
4. A Screening and Baseline visit Clinician-Administered Inventory of Depressive Symptomatology Questionnaire (IDS-C30) score ≥ 25.
5. Screening visit high-sensitivity C-reactive protein (CRP) concentration ≤ 5 mg/L (based on evidence that cytokine antagonism has an independent antidepressant effect in depressed patients with elevated CRP above this cut-off).

Exclusion Criteria:

1. Any of the following medical conditions:

   * cardiovascular disease (other than controlled hypertension)
   * seizure disorder, history of cerebrovascular accident (CVA) or other serious neurological condition (e.g., Parkinson's disease, multiple sclerosis, seizure disorder [except childhood febrile seizures], dementia or delirium)
   * presence or history of neoplasia (other than resected non-melanotic skin cancer)
   * endocrinopathies (diabetes mellitus types I and II, Cushing's disease, Addison's disease)
   * active autoimmune disease (e.g., rheumatoid arthritis, Hashimoto's thyroiditis, inflammatory bowel disease)
   * chronic infection (e.g., hepatitis B or C or human immunodeficiency virus [HIV] infection)
   * acute kidney injury or Chronic Kidney Disease
   * any history of or current diagnosis of thrombosis or thrombophilia; if it is unclear whether a subject has received this diagnosis, a signed release will be obtained to contact the subject's treating physician and obtain accurate diagnostic information. Depending on the recommendation of the treating physician, the subject may undergo appropriate testing with the treating physician to verify the diagnosis, and if the tests produce negative findings, the subject may be allowed to enter the study.
   * any history of recurrent or recurring HSV (Herpes simplex)
   * any active enclosed infection (e.g., dental abscess, joint infection)
   * hemophilia or other cause for excessive bleeding (e.g., platelet disorder)
   * fever (Temp > 99) of unknown origin at the time of screen
   * laboratory evidence of undiagnosed hypothyroidism or any change in treatment for hypothyroidism in the 3 months prior to screening.
   * significant electrocardiogram abnormalities
   * plan to receive surgery or medical procedure during the study
   * those with impaired sensation (e.g. diabetic polyneuropathy)
   * those with a deteriorated ability to express themselves
   * those in whom irradiating cold tissue, tissue badly supplied with blood or an area with low subcutaneous tissue (e.g. tibial border)
2. Any other medical condition that in the judgment of the PI would increase the risk of study participation or introduce excessive physiological variance into the study population
3. A positive score to C-SSRS items 4 or 5 is OR a suicide attempt in the past 12 months
4. Morbid obesity and/or body shape that might increase the risk of cutaneous burning from the Heckel HT3000 hyperthermia device (because of truncal skin being too close to the infrared lights defined as 3 inches or less)
5. Breast implants (because these increase the risk of burning)
6. Known hypersensitivity to hyperthermia and/or infrared exposure
7. Evidence of sunburn at time of treatment intervention
8. Use of any medication that might impact thermoregulatory capacity within 5 days of receiving WBH treatment, including: stimulants, diuretics, barbiturates, beta-blockers, antipsychotic agents, anti-cholinergic agents or chronic use of antihistamines, aspirin (other than low-dose ASA for prophylactic purposes), non-steroidal anti-inflammatory drugs (NSAIDs), systemic corticosteroids, cytokine antagonists
9. Use of any other medication that in the judgment of the PI would increase risk of study participation or introduce excessive variance into physiological or behavioral responses to WBH
10. Breastfeeding or pregnant women, women intending to become pregnant within 6 months of the screening visit, or sexually-active women of child bearing potential who are not using a medical accepted means of contraception (defined as oral contraceptive pill or implant, condom, diaphragm, IUD, status-post tubal ligation, or partner with vasectomy)
11. Any of the following exclusionary conditions for treatment with tocilizumab:

    * Taking immunosuppressive drugs including but not limited to:

      * Disease-modifying anti-rheumatic drugs (DMARDs) such as methotrexate
      * Corticosteroids such as prednisone
      * Monoclonal antibodies such as anti-CD20 monoclonal antibodies
    * Taking selective co-stimulation modulators
    * Regularly taking nonsteroid anti-inflammatory drugs (NSAIDs) or COX-2 inhibitors in the 24 hours prior to WBH treatment and/or biomarker assessment
    * Absolute neutrophil count (ANC) below 2000 per mm3 or a history of neutropenia
    * Platelet count below 100,000 per mm3 or a history of thrombocytopenia
    * Elevated ALT or AST levels above 1.5 times the upper limit of normal (ULN)
    * Known hypersensitivity to tocilizumab or other ingredients in ACTEMRA
    * History of tuberculosis (TB), past exposure to TB, positive TB test result, residence or travel to areas of endemic TB or endemic mycoses within previous 6 months, meets TB risk factors after evaluation
    * History of having received the Bacillus Calmette-Guérin (BCG) vaccine
    * Has an underlying condition that may predispose them to infection (e.g., HIV, autoimmune disorders, on chemotherapy, etc)
    * Has a history of or an increased risk for gastrointestinal perforation such as a history of diverticulitis, stomach or intestinal ulcers or abdominal pain that does not go away
    * History of demyelinating disorders such as multiple sclerosis or chronic inflammatory demyelinating polyneuropathy
    * Have received a live vaccination in the one month prior to the scheduled administration of tocilizumab
12. A lifetime history of any Psychotic Disorder, bipolar I or II disorder, anorexia nervosa
13. Meeting DSM-5 criteria at screening for current obsessive compulsive disorder or bulimia nervosa.
14. Patients who have failed to respond during the course of their current major depressive episode to >4 adequate antidepressant trials, defined as six weeks or more of treatment with the FDA-defined minimally effective dose, as assessed by the ATRQ.
15. A concurrent anxiety disorder (e.g., obsessive compulsive disorder, panic disorder, posttraumatic stress disorder) that appears to be an individual's primary clinical problem (with the result that depressive symptoms are judged to either result from this primary condition or to be secondary to it)
16. A concurrent personality disorder (e.g., borderline personality disorder, narcissistic personality disorder, histrionic personality disorder) that appears to be an individual's primary clinical problem (with the result that depressive symptoms are judged to either result from this primary condition or to be secondary to it)
17. Meets criteria for any substance use disorder in 3 months previous to screening (except for nicotine or caffeine use disorder)
18. Lifetime history of antisocial personality disorder
19. Use of antidepressant or other psychotropic medications (other than benzodiazepine or non-benzodiazepine sleeping aids, e.g., zolpidem at a stable dose for at least 4 weeks) within 4 weeks of screening (8 weeks for fluoxetine due to its extended half-life)
20. Participation in ongoing psychotherapy unless it has been stable for at least 3 months and individual has not improved (i.e., still meets criteria for MDD per MINI)
21. Commencement of any psychotropic or psychotherapeutic intervention between screening and study completion
22. A score of 4 or 5 on the Columbia Suicide Rating Scale (C-SSRS), consistent with active suicidal ideation with specific plan and intent, or suicide attempt within 12 months of screening per self-report
23. Claustrophobia of sufficient severity to interfere with ability to enter/remain in Heckel HT3000 device

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2026-12-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Inventory of Depressive Symptomatology Self-Report (IDS-SR) | Week 0 (Visit 2) to Week 1 (visit 3) [approximately 7 days]
  The IDS-SR is a self-administered questionnaire assessing depressive severity. 30 questions focus on depressive symptoms experienced over the past 7 days. Each question is scored from 0-3, for a total minimum score of 0 and a total maximum score of 84 (appetite and weight items are split into two questions each, one for increase and one decrease, but counted once only, so there are effectively 28 items). Higher scores indicate more severe depression. Ranges correspond to depressive severity as follows: 0-13 = no or minimal depression; 14-25 = mild depression; 26-38 = moderate depression; 39-48 = severe depression; 49-84 = very severe depression. A decrease of 50% or more in the score is considered to be a response to treatment, while a final score of 11 or less is considered remission. Primary study outcomes will be between-group differences (tocilizumab vs. placebo) in total IDS-SR score change from Week 0 (Visit 2) to Week 1 (visit 3).

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Janssen CW, Lowry CA, Mehl MR, Allen JJ, Kelly KL, Gartner DE, Medrano A, Begay TK, Rentscher K, White JJ, Fridman A, Roberts LJ, Robbins ML, Hanusch KU, Cole SP, Raison CL. Whole-Body Hyperthermia for the Treatment of Major Depressive Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2016 Aug 1;73(8):789-95. doi: 10.1001/jamapsychiatry.2016.1031. PMID 27172277
- [Background] Hanusch KU, Janssen CH, Billheimer D, Jenkins I, Spurgeon E, Lowry CA, Raison CL. Whole-body hyperthermia for the treatment of major depression: associations with thermoregulatory cooling. Am J Psychiatry. 2013 Jul;170(7):802-4. doi: 10.1176/appi.ajp.2013.12111395. No abstract available. PMID 23820835
- [Background] Hale MW, Lukkes JL, Dady KF, Kelly KJ, Paul ED, Smith DG, Raison CL, Lowry CA. Whole-body hyperthermia and a subthreshold dose of citalopram act synergistically to induce antidepressant-like behavioral responses in adolescent rats. Prog Neuropsychopharmacol Biol Psychiatry. 2017 Oct 3;79(Pt B):162-168. doi: 10.1016/j.pnpbp.2017.06.006. Epub 2017 Jun 12. PMID 28619470